CLINICAL TRIAL: NCT02616315
Title: A Randomized, Double-Blind, Phase 4 Study to Evaluate the Efficacy of Naltrexone HCl/Bupropion HCl Extended Release Versus Placebo for Treatment of Weight Regain in Patients Post Bariatric Surgery
Brief Title: Efficacy of Naltrexone HCl/Bupropion HCl Extended Release Versus Placebo for Treatment of Weight Regain in Participants Post Bariatric Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NaltrexBuprop-4004; U1111-1168-9817 (Registry Identifier: WHO)
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Weight Regain Post Bariatric Surgery
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Placebo (Placebo Comparator): Naltrexone hydrochloride (HCl)/bupropion hydrochloride (HCl) placebo-matching tablet, orally, 1 tablet in the AM, daily, during Week 1, followed by naltrexone HCl/bupropion HCl placebo-matching tablets, orally, 1 tablet in the AM and 1 in the PM, during Week 2, followed by naltrexone HCl/bupropion HCl placebo-matching tablets, orally, 2 tablets in the AM and 1 in the PM, during Week 3, followed by naltrexone HCl/bupropion HCl placebo-matching tablets, orally, 2 tablets in the AM and 2 in the PM, in Week 4 through Week 49. Participants must be re-titrated if off treatment for ≥1 week (≥7 days).
  Interventions: Drug: Naltrexone HCl/Bupropion HCl Placebo
- Group B: Naltrexone HCl/Bupropion HCl (Experimental): Naltrexone HCl 8 mg/bupropion HCl 90 mg, tablet, orally, 1 tablet in the AM, daily, during Week 1, followed by naltrexone HCl 8 mg/bupropion HCl 90 mg, tablets, orally, 1 tablet in the AM and 1 in the PM, during Week 2, followed by naltrexone HCl 8 mg/bupropion HCl 90 mg, tablets, orally, 2 tablets in the AM and 1 in the PM, during Week 3, followed by naltrexone HCl 8 mg/bupropion HCl 90 mg, tablets, orally, 2 tablets in the AM and 2 in the PM, in Week 4 through Week 49. Participants must be re-titrated if off treatment for ≥1 week (≥7 days).
  Interventions: Drug: Naltrexone HCl/Bupropion HCl

INTERVENTIONS:
Drug: Naltrexone HCl/Bupropion HCl Placebo — Naltrexone/bupropion placebo-matching tablets
  Arms: Group A: Placebo
Drug: Naltrexone HCl/Bupropion HCl — Naltrexone HCl 8 mg/bupropion HCl 90 mg tablets
  Arms: Group B: Naltrexone HCl/Bupropion HCl

SUMMARY:
The purpose of this study is to determine the effect of naltrexone hydrochloride(HCL) and bupropion hydrochloride extended release combination (NB) compared with placebo on weight loss in obese participants post bariatric surgery.

DETAILED DESCRIPTION:
The drug being tested in this study is called naltrexone hydrochloride/bupropion hydrochloride (NB). NB is being tested to determine its effect on weight loss in obese participants post bariatric surgery.

The study will enroll approximately 60 participants. Participants will be randomly assigned to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Naltrexone HCl 32 mg/bupropion HCl 360 mg extended-release tablet
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants will start on 1 tablet a day and will increase their dose by 1 tablet per week for 4 weeks to reach the optimal dose.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 59 weeks maximum. Participants will make multiple visits to the clinic, plus a final visit 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is female or male and aged 18 to 65 years, inclusive.
4. Is at least 2 years post Roux-en-Y Gastric Bypass (RYGB) procedure for treatment of severe obesity prior to screening.
5. Has achieved an initial weight loss of ≥20% of their preoperative body weight, and has regained ≥10% of the total weight lost.
6. Has a body mass index (BMI) (weight [kg]/[height {m}]^2) ≥30 kg/m^2.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after the last dose of study drug.
8. Is able to speak and read English.

Exclusion Criteria:

1. Has obesity of known endocrine origin (eg, untreated hypothyroidism, Cushing's syndrome) or of genetic origin.
2. Is currently using other bupropion- or naltrexone-containing products or has a history of hypersensitivity or allergies to naltrexone or bupropion.
3. Has a history of cancer that has been in remission for <5 years prior to screening. A history of basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin is allowed.
4. Has a history of Type 1 or current type 2 diabetes mellitus (T2DM) diagnosis.
5. Has had a myocardial infarction within 6 months prior to screening.
6. Has a history of Class III or IV congestive heart failure, as per the New York Heart Association functional classification.
7. Has a history of angina pectoris Grade III or IV, as per the Canadian Cardiovascular Society grading scheme.
8. Has a clinical history of strokes, including ischemic and hemorrhagic strokes.
9. Has a history (within the last 20 years) of seizures, cranial trauma, active bulimia, anorexia nervosa, or other conditions that predispose the participant to seizures.
10. Has, in the judgment of the investigator, any clinically significant electrocardiogram (ECG), laboratory, hematology, physical examination, medical history, or urinalysis finding that should prohibit participation in the study.
11. Has uncontrolled hypertension defined as blood pressure (BP) ≥145/95 mm Hg at screening. BP will be measured on 2 separate occasions with an approximate 30-minute interval between measurements at the screening visit.
12. Has a thyrotropin (thyroid stimulating hormone -TSH) value outside the normal range at the screening visit; unless there is a normal triiodothyronine (T3) value.
13. Had initiation or alteration of dose of antihypertensive or lipid-lowering agents within 4 weeks prior to screening.
14. Used prescribed or over-the-counter drugs intended for weight loss, or participated in a weight loss program other than standard of care for a post bariatric population, within 3 months prior to randomization.
15. Has prior or planned surgical or device intervention for obesity except for the required RYGB Surgery.
16. Has a history or current diagnosis of angle-closure glaucoma.
17. Is experiencing post bariatric dumping syndrome that may impact the conduct or outcome of the study as determined by the investigator.
18. Has moderate or severe renal impairment (end-stage renal disease) defined as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m^2, using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI).
19. Has a clinical history of hepatic impairment or current documented aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN) at the screening visit.
20. Has glycosylated hemoglobin (HbA1c) ≥6.5% at Screening Visit.
21. Has current known infection with human immunodeficiency virus (HIV) or hepatitis (documentation of no detectable virus is required for participants with a past infection of hepatitis B or C).
22. Is undergoing an abrupt discontinuation of alcohol, benzodiazepines, barbiturates, or antiepileptic drugs.
23. Is a chronic user or has a positive screen for opioids.
24. Has a hemoglobin of ≤10 g/100 mL at the screening visit.
25. Has a history of serious psychiatric illness such as:

    * A Patient Health Questionnaire (PHQ)-9 score ≥10 at the screening visit.
    * Bipolar disorder.
    * Schizophrenia.
    * Severe personality disorder (eg, borderline or antisocial).
    * Major depressive disorder.
    * Recent (previous 6 months) suicide attempt.
    * Other psychosis.
26. If female, the participant is pregnant or trying to become pregnant, currently breast-feeding, or of childbearing potential (including perimenopausal women who have had a menstrual period within 1 year) and not willing to practice birth control from signing of informed consent throughout the duration of the study and for 12 weeks after the last dose of study drug.
27. Has received any investigational compound within 30 days prior to the first dose of study medication.
28. Has received Contrave in a previous clinical study or as a therapeutic agent.
29. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
30. Is required to take excluded medications.
31. Participant is enrolled in any other interventional study at the time of Screening and during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight at Week 26 | Baseline and Week 26

SECONDARY OUTCOMES:
Percent Change from Baseline in Body Weight at Week 52 | Baseline and Week 52
Percentage of Participants Achieving a Loss of at Least 2%, 5%, or 10% of Baseline Body Weight at Weeks 26 and 52 | Baseline and Weeks 26 and 52
Changes from Baseline on Obesity-Associated Cardiovascular Risk Factors at Weeks 26 and 52 | Baseline and Weeks 26 and 52
  Obesity-associated cardiovascular risk factors, including serum triglycerides, high density lipoprotein (HDL), and low density lipoprotein (LDL) cholesterol, and waist circumference.
Change from Baseline in Fasting Glucose Levels at Weeks 26 and 52 | Baseline and Weeks 26 and 52
Change from Baseline in and Glycosylated Hemoglobin (HbA1c) Levels at Weeks 26 and 52 | Baseline and Weeks 26 and 52
Change from Baseline in Vital Signs at Weeks 26 and 52 | Baseline and Weeks 26 and 52
  Vital signs include systolic and diastolic blood pressure [BP] and heart rate.
Change from Baseline in Quality of Life as Measured by the Impact of Weight on Quality of Life Questionnaire - Lite Version (IWQOL-Lite) at Weeks 26 and 52 | Baseline and Weeks 26 and 52
  The IWQOL-Lite, is a validated 31-item, self -reported, obesity-specific measure of health-related quality of life that consists of a total score and scores on each of 5 scales (physical function, self-esteem, sexual life, public distress, and work) that exhibits strong psychometric properties. Participants rate items within the scales as: 5=always true, 4=usually true, 3=sometimes true, 2=rarely true, or 1=never true. Scale scores are obtained by adding item scores, and the total score is obtained by adding scale scores. Higher scores indicate poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director US Medical Affairs, Study Director — Takeda
Locations (2):
- United States (2):
  - Chicago, Illinois
  - Boston, Massachusetts